CLINICAL TRIAL: NCT01641211
Title: Using MEDUCATION to Improve Asthma Medication Device Technique
Brief Title: ENLaCE Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Delesha Carpenter, PhD, MSPH, Research Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-1008
Record Dates: First submitted 2012-07-09; First posted 2012-07-16 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video intervention (Experimental): Group that will watch the Meducation inhaler device technique videos.
  Interventions: Behavioral: Meducation device technique video
- Control (Other): This group will watch a nutrition video.
  Interventions: Other: Nutrition video

INTERVENTIONS:
Behavioral: Meducation device technique video — 2-minute video that displays proper inhaler, diskus, and turbuhaler technique. The video will only be watched once at the medical visit. Children in this group will be given a wallet card so they can access the video via the Internet after leaving the asthma clinic.
  Arms: Video intervention
Other: Nutrition video — Children in this group will watch a 2-minute nutrition video.
  Arms: Control

SUMMARY:
This is a feasibility study to determine whether the Expanding Networks for Latinos through Community Engagement (ENLaCE) can be used to recruit Latino children into a randomized, controlled trial (RCT) to improve their asthma medication device technique. Children will be recruited from two pediatric ENLaCE clinics in Greensboro and randomly assigned to watch device technique videos (experimental group; n=50) or a nutrition video (control group, n=50) in Spanish or English after a regularly-scheduled medical visit. Children's device technique will be assessed before and after the visit. Process evaluation data will also be collected. The investigators hypothesize that children in the intervention group will have better device technique post-intervention than the control group.

DETAILED DESCRIPTION:
Asthma affects almost 10% of children and is the most common health condition reported by North Carolina public schools. Latino children have higher rates of uncontrolled asthma and more asthma-related emergency department visits than their White counterparts. No studies have evaluated Latino children's asthma device technique; poor technique can compromise medication delivery to the lungs.

The TraCS engagement core has spent the last 18 months developing the Expanding Networks for Latinos through Community Engagement (ENLaCE) network, which is comprised of over 15 organizations in the Greensboro area. The core would now like to conduct a feasibility study to determine whether ENLaCE can be used to recruit Latino children into a randomized, controlled trial (RCT) to improve their asthma medication device technique. This would be the first assessment of whether ENLaCE can be used to recruit patients.

MEDUCATION, an NIH-funded project developed by Polyglot Systems, Inc., has developed asthma device technique videos in Spanish and English. The member groups of ENLaCE believe the MEDUCATION videos are highly relevant for the Greensboro Latino community. Children will be recruited from two pediatric ENLaCE clinics in Greensboro and randomly assigned to watch device technique videos (experimental group; n=50) or a nutrition video (control group, n=50) in Spanish or English after a regularly-scheduled medical visit. Children's device technique will be assessed before and after the visit. Process evaluation data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

Children will be eligible if they:

* are ages 8 through 16 years,
* are able to speak English or Spanish,
* can read the assent form,
* are present at the visit with an adult caregiver (parent or legal guardian) who can speak English or Spanish and who is at least 18 years of age,
* have mild, moderate, or severe persistent asthma, and
* are present for an asthma-related visit (either acute or scheduled).

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in inhaler, turbuhaler, and diskus technique | Baseline and 1-month follow-up
  Children will demonstrate how they use their metered-dose inhalers, turbuhalers, and diskuses using empty devices. The research assistant will record the number of steps performed correctly. Correct use of inhalers, diskuses, and turbuhalers will be measured as continuous variables.

SECONDARY OUTCOMES:
Child inhaler self-efficacy | Baseline and 1-month follow-up
  Child inhaler self-efficacy will be measured as a continuous variable using 1 item from the Bursch asthma management self-efficacy measure, "How sure are you that you can use your inhaler correctly?"
Asthma Control | Baseline and 1-month follow-up
  The Asthma Control Test is a 5-item questionnaire assessing asthma symptoms, use of rescue medications, and the effect of asthma on daily functioning. Scores range from 5 (poor control) to 25 (complete control). Studies show that the Asthma Control Test is reliable, valid, and responsive to temporal changes in asthma control.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomasville Pediatrics, Thomasville, North Carolina, United States

REFERENCES:
- [Derived] Carpenter DM, Lee C, Blalock SJ, Weaver M, Reuland D, Coyne-Beasley T, Mooneyham R, Loughlin C, Geryk LL, Sleath BL. Using videos to teach children inhaler technique: a pilot randomized controlled trial. J Asthma. 2015 Feb;52(1):81-7. doi: 10.3109/02770903.2014.944983. Epub 2014 Jul 31. PMID 25025548